CLINICAL TRIAL: NCT06469866
Title: Effect of Deep Neuromuscular Block on the Quality of Recovery After Laparoscopic Hysterectomy
Brief Title: Deep Neuromuscular Block Affect the Quality of Recovery After Laparoscopic Hysterectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anqing Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: xuzhang520
Record Dates: First submitted 2024-06-11; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Neuromuscular Blockade; Laparoscopy
Keywords: Neuromuscular block; Recovery; Laparoscopic hysterectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-pressure pneumoperitoneum (LPP) with deep NMB affect quality of recovery (Experimental): low-pressure pneumoperitoneum (LPP) with deep NMB.
  Interventions: Device: low-pressure pneumoperitoneum; Device: standard-pressure pneumoperitoneum
- standard-pressure pneumoperitoneum (SPP) with moderate NMB affect quality of recovery (Experimental): standard-pressure pneumoperitoneum (SPP) with moderate NMB.
  Interventions: Device: low-pressure pneumoperitoneum; Device: standard-pressure pneumoperitoneum

INTERVENTIONS:
Device: low-pressure pneumoperitoneum — low-pressure pneumoperitoneum (LPP) with deep NMB.
Device: standard-pressure pneumoperitoneum — standard-pressure pneumoperitoneum (SPP) with moderate NMB.

SUMMARY:
BACKGROUND: Some studies have revealed that deep neuromuscular block (NMB) improve surgical conditions and alleviated postoperative pain compared with moderate NMB. The present study investigated deep NMB could improve the quality of recovery after laparoscopic hysterectomy

METHODS: seventy-two women with elective laparoscopic hysterectomy were randomly divided into 2 groups: Patients in group A received low-pressure pneumoperitoneum (LPP), which was set at 8-10 mmHg with deep NMB. Patients in group B received standard-pressure pneumoperitoneum (SPP), which was set at 12-14 mmHg with moderate NMB. Primary outcome was the quality of recovery (QoR-15) at 1 day after sugery. The secondary outcomes included postoperative pain, surgical condition, incidence of shoulder pain, the incidence of rescue analgesic drug use, cumulative dose of analgesics, time of first flatus, post-operative nausea and vomiting, time of tracheal tube removal.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status Ⅰ- Ⅲ
* Scheduled for elective laparoscopic hysterectomy

Exclusion Criteria:

* Inability to give informed consent
* BMI >35
* Renal or hepatic insufficiency
* History of preoperative psychiatric
* Previous surgery at procedure site
* Neuromuscular disease, pregnancy, and contraindications to study medications.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-06-25 (Estimated); Primary Completion 2024-11-25 (Estimated); Study Completion 2024-11-25 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery | 1 day after operation
  Primary outcome measure was the quality of recovery at 1 day after surgery. Quality of recovery-15 scale was used to assess the quality of recovery after operation. A higher score of quality of recovery-15 scale indicates a better quality of recovery after surgery

SECONDARY OUTCOMES:
Shoulder pain | The first 24 hours after operation
  Secondary Outcome Measure was the incidence of shoulder pain
Postoperative nausea and vomiting | The first 24 hours after operation
  Secondary Outcome Measure was the incidence of postoperative nausea and vomiting. PONV score was evaluated verbally with a descriptive scale (0 = None, 1 = Mild Nausea, 2 = Moderate Nausea, 3 = One Vomiting, 4 = Multiple Vomiting).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anqing Munucipal Hospital Anesthesiology, Anqing, Anhui, China